CLINICAL TRIAL: NCT05600829
Title: A Behavioural Weight Loss Intervention Delivered in Cardiac Rehabilitation for Patients With Atrial Fibrillation and Obesity: The BeWEL IN CR-AF Study
Brief Title: A Behavioural Weight Loss Intervention Delivered in Cardiac Rehabilitation for Patients With Atrial Fibrillation and Obesity
Acronym: BeWEL IN CR-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Tavis S. Campbell, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB22-0976
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation; Obesity
MeSH Terms: conditions — Atrial Fibrillation; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients participate in a traditional 12-week outpatient CR program with added weekly behavioural weight loss classes.
  Interventions: Behavioral: BWLT+CR
- Control (Other): Patients participate in a traditional 12-week outpatient CR program.
  Interventions: Behavioral: CR-Only

INTERVENTIONS:
Behavioral: BWLT+CR — Patients will attend twelve 2-hour group-based weekly sessions (over Zoom) in addition to their twice-weekly CR exercise sessions, followed by biweekly follow-up sessions alternating between individual phone-based sessions with a facilitator, and group-based sessions for an additional 12 weeks. The empirically validated ASPIRE BWLT was recently adapted for an AF population with obesity. Briefly, the BWLT was modified to incorporate education and practical strategies requested by patients, including AF risk factor management, pathophysiology, medications, and disease course; exercising with AF; and coping with difficult emotions regarding AF. Weekly treatment goals focus on nutrition and moderate calorie reduction while emphasizing adherence to an individualized CR exercise prescription. The BWLT program will be delivered by senior clinical psychology PhD students and supervised by a registered Clinical Health Psychologist.
  Arms: Intervention
Behavioral: CR-Only — The CR program consists of education, medication management, risk factor modification and 12 weeks of twice-weekly supervised cardiovascular exercise sessions. Patients with AF undergo a symptom-limited graded exercise stress test at intake, 12-weeks, 24-weeks, and 1-year post-randomization, where cardiorespiratory fitness (i.e., peak metabolic equivalents [METS]) and cardiometabolic risk factors (blood pressure, blood lipid profile, BMI, waist circumference, depression and anxiety symptoms, tobacco use, and exercise volume) are assessed.
  Arms: Control

SUMMARY:
One-in-four Canadians will be diagnosed with an abnormal heart rhythm called atrial fibrillation (AF) in their lifetime. This is expected to double by 2050, owing to an aging population and increased age- and health behaviour-associated AF risk factors (e.g., poor cardiorespiratory fitness, Type II diabetes, hypertension, and obesity). AF is associated with an increased risk of severe health outcomes including stroke, heart failure, dementia, and death. Nearly three-quarters of people with AF also have obesity (excess body weight). According to research, people with obesity that lose approximately 10% of their body weight can experience relief from uncomfortable AF symptoms. Losing weight may even help people return to a normal heart rhythm.

Cardiac rehabilitation (CR) is a proven way to help people with heart disease live longer, healthier lives. So far, research has not shown whether CR helps improve the abnormal heart rhythms seen in AF. This may be because CR programs usually do not offer specific help with weight management. Therefore, adding behavioural weight-loss treatment (BWLT; group classes to change thoughts and behaviours to encourage weight loss) to CR programs may help people with AF and obesity experience relief from their symptoms.

This randomized controlled trial will assess whether the combination of an AF-specific 'small changes' BWLT and traditional CR results in a greater proportion of patients with AF and obesity achieving ≥ 10% body weight loss compared to patients who receive standard care (traditional CR alone). Traditional CR consists of participating in exercise sessions, supervised by health professionals, twice per week for 12 weeks. In addition to traditional CR, patients that are randomized to receive BWLT will attend 12 weekly online group therapy classes to learn strategies from psychology to help encourage weight loss. The investigators will collect data pertaining to weight, AF burden, physical activity, and disease-specific and generic patient-reported outcomes. This information will determine if taking CR+BWLT helps patients with weight loss and AF symptoms. Further, it will help efforts to provide effective treatment to patients with AF to help participants lose weight and reduce or eliminate AF symptoms.

DETAILED DESCRIPTION:
Background: One-in-four Canadians will develop atrial fibrillation (AF), increasing risk of heart failure and stroke. Obesity (i.e., BMI ≥30 kg/m2) represents a strong, independent risk factor for increased incidence and severity of AF. Weight loss reduces AF symptom burden, and patients with obesity who lose ≥10% of their body weight may achieve AF regression/remission. Cardiac rehabilitation (CR) improves AF risk factors including hypertension and cardiorespiratory fitness (CRF), yet the efficacy of CR for reducing AF symptom burden is not established. CR rarely includes targeted obesity management and, on average, has a negligible impact on BMI. Adding behavioural weight-loss treatment (BWLT) to traditional CR may therefore enhance weight loss and lead to improvements in AF prognosis, symptoms, and health-related quality-of-life (HRQOL) in patients with AF and obesity.

Given the high prevalence of obesity among individuals with AF, and its detrimental effect on AF burden and outcomes, there is a critical need for interventions that can support weight-loss-promoting behaviours and can be integrated into routine clinical care for AF. CR programs are available in all major Canadian cities and have a proven track-record of achieving clinically-relevant improvements in important AF risk factors including hypertension, lipid profile, and exercise capacity. Therefore, CR represents an ideal setting to promote risk factor management for patients with AF. Yet, because traditional CR does not produce meaningful weight loss there is a clear gap in the ability of current CR programming to meet the needs of a growing population of individuals with AF and obesity. The addition of a novel BWLT component to CR is needed to bridge this gap and provide the appropriate treatment regimen of comprehensive risk factor management, exercise, and weight loss to achieve optimal AF outcomes.

The primary aim is to: Assess whether the combination of an AF-specific 'small changes' BWLT and traditional CR results in a greater proportion of patients with AF and obesity achieving ≥ 10% body weight loss compared to patients who receive standard care (traditional CR alone).

The secondary aims of the proposed study are to evaluate the impact of BWLT+CR on: 1) mean % weight loss of controls vs. intervention group; 2) AF burden; 3) self-reported AF symptom burden; 4) disease-specific and generic patient-reported outcome measures (e.g., AF- and health-related quality-of-life [HRQoL]; psychological distress); and 5) exercise volume measured in weekly steps.

Hypotheses:

The primary study hypothesis is that patients in the BWLT+CR group will be more likely to achieve ≥10% weight loss at 12 months post-randomization relative to the CR-only group.

Secondary hypotheses are that: patients in the BWLT+CR group will experience greater improvements in AF burden, AF self-reported symptom burden, increased HRQoL, decreased psychological distress, and increased leisure-time exercise and CR exercise session attendance relative to the CR-only group.

Study design:

Design and Procedure. Patients will be assessed for eligibility at TotalCardiology Rehabilitation (TCR). Eligible patients who consent to participate will be enrolled into the CR program and randomized to either the BWLT+CR or CR-only group. Prior to randomization, patients will complete a questionnaire battery including socio-demographic variables (age, sex, ethnicity, income, education), self-reported weight and height to establish BMI, and validated questionnaires assessing AF symptom burden, AF-related quality-of-life, general HRQOL, and psychological distress at baseline (T1). Patients will be re-administered the test battery following the 12-week BWLT+CR program, or 12 weeks of the CR-only program (T2). (Note: T2 measures will be administered even if the patient is still completing their remaining CR exercise sessions. CR completion/adherence will be determined after patients have completed their 12-week exercise program). The test battery will be administered for a final time approximately 24 weeks post-randomization. Weight loss from baseline to 52-weeks will be calculated and converted to a percentage of initial body weight at baseline. Clinical variables (e.g., CRF from graded exercise tests; blood pressure, lipids) will be obtained by TCR chart review.

Recruitment. Patients will be recruited in two ways: (1) directly from TotalCardiology Rehabilitation using referrals from Dr. Wilton and TCR clinic staff, and (2) from an existing database of patients who participated in the Part I qualitative study and Part II acceptability study that provided consent to be contacted about future studies. The recruitment period will be from October 2022 to April 2024. Equal numbers of men and women will be recruited. AF clinic patients who are both (a) eligible for the CR program and (b) eligible for the proposed study will be identified by Dr. Wilton and/or TCR clinic staff. Dr. Wilton/TCR clinic staff will inform patients who meet (a) and (b) criteria about the study and invite them to participate. Interested patients will receive a CR referral and their contact information will be provided to the research coordinator. The research coordinator (B. Valdarchi) will contact patients, provide additional information about the study, and obtain informed consent. The research coordinator will then send an email link to complete baseline questionnaires. Following the completion of the questionnaires, participants will be informed about the group they were randomized to, and scheduled for BWLT groups if needed. Concurrently, patients will be contacted by CR staff to schedule their orientation appointment, as per typical clinic procedures. This recruitment procedure will also apply to patients who previously participated in Part I and II (i.e the qualitative and acceptability studies, respectively). TCR patients who are currently enrolled in CR will also be recruited. A research team member will identify CR patients who have consented to be approached about research and who are eligible for inclusion by reviewing patient chart data. An RA will contact patients by telephone to review study procedures and obtain patients' informed consent.

Sample Size/Analysis. Analysis will be by intention to treat. Conservatively assuming a 5% success rate in the control group and a 30% success rate in the intervention group, 78 patients (39 per group) will provide 80% power to detect a difference using a two-sided independent test of proportions with a 5% significance level. The investigators estimate loss to follow-up and drop-outs of 20% and 10% respectively, therefore 120 patients will be recruited in total (60 per group). The primary analysis will compare the proportion in each group achieving ≥10% weight loss between baseline and 52 weeks post-randomization. A secondary per-protocol analysis will be performed including only participants who complete at least the initial 12-weeks of the BWLT. AF burden will be calculated as a % of total ECG tracings and compared between treatment and controls. Self-reported secondary outcomes will be evaluated using linear mixed modelling.

ELIGIBILITY:
Inclusion Criteria:

* Adults of age ≥18 years
* Symptomatic paroxysmal or persistent atrial fibrillation or atrial flutter
* Classified as obese (BMI ≥30 kg/m2)
* Have a sedentary lifestyle (not currently meeting basic physical activity targets of ≥150 minutes/week)
* Ability to speak and write in English
* Willingness to be referred to a behavioural weight loss treatment (BWLT)
* At least one of the following: obstructive sleep apnea, diabetes, hypertension, heart failure, dyslipidemia, CAD, peripheral artery, or cerebrovascular disease.

Exclusion Criteria:

* Longstanding-persistent (defined as ≥ 3 years continuous AF) or permanent AF
* Uncontrolled coronary artery disease
* Completed a CR program within the previous year
* Currently enrolled in a structured behavioural weight loss program
* Currently scheduled to receive catheter ablation in AF
* Currently taking GLP-1 receptor agonist or
* Received bariatric surgery in the previous year prior to enrollment OR scheduled for bariatric surgery during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving ≥10% body weight change | Baseline, 52 weeks
  Assessed by dividing the number of kilograms at 52 weeks by the initial (T1) kg and multiplying by 100%.

SECONDARY OUTCOMES:
Total Weight Loss | Baseline, 12 weeks, 24 weeks, 52 weeks
  Assessed by dividing the number of kilograms lost at 52 weeks by initial (T1) kg, multiplying by 100% and comparing across conditions. Weight used for outcome analyses will be recorded by TCR staff at the T1 (baseline) T2, (12 weeks), T3 (24 weeks) and T4 (52 week) follow up visits.
AF Burden | 12 weeks, 24 weeks, 52 weeks
  Assessed by daily ECG monitoring with the AliveCor™ KardiaMobile EKG device. Patients in both groups will record 30sec ECGs twice daily. Tracings will be sorted by the AliveCor AI software and abnormal tracings will be reviewed by cardiology residents at the University of Calgary to identify tracings with AF. Total AF burden will be calculated as the percentage of all ECG tracings showing AF from weeks 12-52, to allow for latency of intervention effect on AF pathophysiology. Multiple imputation will be used to handle missing ECG data. A biostatistician will be consulted to assist with statistical procedures.
AF Symptom Burden | Baseline, 12 weeks, 24 weeks
  University of Toronto AF Symptoms Severity Scale (AFSS) - The AFSS assesses subjective and objective AF disease burden across four domains: AF burden (frequency, duration, and severity of AF episodes); global well being (visual analogue scale where patients rate their life from "worst" to "best" 1-10).
AF-related Quality of Life | Baseline, 12 weeks, 24 weeks
  Atrial Fibrillation Effect on Quality-of-Life Questionnaire (AFEQT) - The AFEQT is a 20-item self-report questionnaire assessing impact of AF across four QOL domains: symptoms, daily activities, treatment concern, and treatment satisfaction. A large (6-centre) prospective validation study indicates the AFEQT has high (> 0.88) internal consistency, and is sensitive to intervention effects (i.e., scores increased 3-month post-ablation). Lower AFEQT scores are associated with increased AF severity.
Symptoms of Psychological Distress | Baseline, 12 weeks, 24 weeks
  Hospital Anxiety and Depression Scale (HADS) - The HADS is a 14-item self-report questionnaire that measures anxiety (HADS-A) and depression (HADS-D). It has well-established cut-offs for minimal, mild, moderate, and severe anxiety and depression symptoms, with higher scores indicating greater psychological distress.
CR Exercise Session Adherence | 12 weeks
  Measured by chart review upon completion of the 12-week exercise program and defined as the # of sessions attended out of 24 sessions.
Weekly Step Counts | 12 weeks, 24 weeks
  Measured using Fitbit fitness trackers. A research assistant will set up individual FitBit accounts and log in weekly to track patients' steps weekly.
Cardiorespiratory Fitness | Baseline, 12 weeks, 24 weeks, 52 weeks
  Assessed by peak metabolic equivalents (METS) from a symptom-limited graded exercise stress test.

CONTACTS AND LOCATIONS:
Overall Officials: Tavis Campbell, PhD, Principal Investigator — University of Calgary
Locations (1):
- Behavioural Medicine Lab, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williamson TM, Rouleau CR, Wilton SB, Valdarchi AB, Moran C, Patel S, Lutes L, Aggarwal SG, Arena R, Campbell TS. A randomized controlled trial of a "Small Changes" behavioral weight loss treatment delivered in cardiac rehabilitation for patients with atrial fibrillation and obesity: study protocol for the BE-WEL in CR-AF study. Trials. 2024 Oct 11;25(1):671. doi: 10.1186/s13063-024-08527-6. PMID 39394158